CLINICAL TRIAL: NCT04094363
Title: CSD190202: A Randomized, Open-Label, Crossover Study to Assess Elements of Abuse Liability for Two Electronic Nicotine Delivery Systems
Brief Title: CSD190202: Study to Assess Elements of Abuse Liability for Two Electronic Nicotine Delivery Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CSD190202
Record Dates: First submitted 2019-09-16; First posted 2019-09-18 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Smoking; Tobacco Smoking; Tobacco Use
MeSH Terms: conditions — Smoking; Tobacco Smoking; Tobacco Use | interventions — HTR3D protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Product usage order ABCD (Experimental): Subjects will use each of the 4 products (ABCD) sequentially for 1 and 1/2 days during a 9 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product usage order BDAC (Experimental): Subjects will use each of the 4 products (BDAC) sequentially for 1 and 1/2 days during a 9 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product usage order CADB (Experimental): Subjects will use each of the 4 products (CADB) sequentially for 1 and 1/2 days during a 9 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D
- Product usage order DCBA (Experimental): Subjects will use each of the 4 products (DCBA) sequentially for 1 and 1/2 days during a 9 day confinement, followed by a 4 hour Test Session.
  Interventions: Other: Product A; Other: Product B; Other: Product C; Other: Product D

INTERVENTIONS:
Other: Product A — Usual Brand, filtered combustible cigarette
Other: Product B — CSD1902-11, an electronic nicotine delivery system
Other: Product C — CSD1902-21, an electronic nicotine delivery system
Other: Product D — 4mg Nicotine gum

SUMMARY:
This is a randomized, open-label, crossover study designed to evaluate elements of abuse liability (AL) including subjective effects, plasma nicotine uptake, and physiological measures during and following ad libitum use of the investigational products (IPs) by healthy subjects.

DETAILED DESCRIPTION:
The study will recruit smokers of combustible cigarettes.

Potential subjects will complete a pre-screening interview and a Screening Visit to assess their eligibility within 45 days prior to enrollment.

Starting on Day 1, eligible smokers will be confined at the clinical site for 9 days. Subjects will participate in four separate Test Sessions for AL assessment, one for each IP. Each Test Session will last for approximately 4 hours during and following IP use. Subjects will be randomized to use one IP in each Test Session: Usual Brand (UB) combustible cigarettes, nicotine gum, and 2 Electronic Nicotine Delivery Systems (ENDS).

For approximately a day and a half prior to each respective Test Session, IP will be dispensed for ad libitum use for product familiarization.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and willing to sign an informed consent form (ICF) and complete questionnaires written in English.
2. Generally healthy male or female, 21 to 60 years of age, inclusive, at the time of consent.
3. Expired breath carbon monoxide level is ≥ 10 ppm and ≤ 100 ppm at Screening.
4. Positive urine cotinine test at Screening.
5. Smokes only combustible, filtered, non-menthol, 83 mm to 100 mm in length.
6. Agrees to smoke same UB combustible cigarette throughout the study period. UB combustible cigarette is defined as the cigarette brand style currently smoked most frequently by the subject.
7. Smokes at least 10 cigarettes per day (on average) and inhales the smoke, for at least 6 months prior to Screening. Brief periods of abstinence due to illness, quit attempt (prior to 30 days of Screening), or clinical study participation (prior to 30 days of Screening) will be allowed at the discretion of the Principal Investigator (PI).
8. Response at Screening to Fagerström Test for Nicotine Dependence (FTND) Question 1 ("How soon after you wake up do you smoke your first cigarette?") is either "Within 5 minutes" or "6-30 minutes."
9. Willing to use UB combustible cigarette, ENDS, and Nicorette gum during the study period.
10. Willing to abstain from tobacco and nicotine use for at least 12 hours prior to each Test Session.
11. Females must be willing to use a form of contraception acceptable to the PI from the time of signing informed consent until End-of-Study.
12. Agrees to in-clinic confinement of 9 days and 8 nights.

Exclusion Criteria:

1. Presence of clinically significant uncontrolled cardiovascular, pulmonary, renal, hepatic, endocrine, gastrointestinal, psychiatric, hematological, neurological disease, or any other concurrent disease or medical condition that, in the opinion of the PI, makes the study subject unsuitable to participate in this clinical study.
2. History, presence of, or clinical laboratory test results indicating diabetes.
3. Systolic blood pressure of > 160 mmHg or a diastolic blood pressure of > 95 mmHg, measured after being seated for five minutes.
4. Weight of ≤ 110 pounds.
5. Hemoglobin level is < 12.5 for females or <13.0 for males g/dL at Screening.
6. Scheduled treatment for asthma currently or within the past consecutive 12 months prior to the Screening Visit. As-needed treatment, such as inhalers, may be included at the PI's discretion pending approval from the Medical Monitor.
7. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
8. Any history of cancer, except for primary cancers of skin such as localized basal cell/squamous cell carcinoma that has been surgically and/or cryogenically removed.
9. Use of an ENDS or other tobacco or nicotine-containing product (e.g., lozenges, moist snuff) within (≤) 30 days prior to Screening.
10. Use of any medication or substance that aids in smoking cessation, including but not limited to any Nicotine Replacement Therapy (NRT) (e.g., nicotine gum, lozenge, patch), varenicline (Chantix®), bupropion (Wellbutrin®, Zyban®), or lobelia extract within (≤) 30 days prior to the signing of informed consent.
11. History or presence of bleeding or clotting disorders.
12. Any use of anticoagulants or aspirin (≥ 325 mg/day).
13. Whole blood donation within 8 weeks (≤ 56 days) prior to the signing of informed consent.
14. Plasma donation within (≤) 7 days prior to the signing of informed consent.
15. Participation in another clinical trial within (≤) 30 days prior to the signing of informed consent. The 30-day window for each subject will be derived from the date of the last study event in the previous study to the time of signing the ICF in the current study.
16. Females who have a positive pregnancy test, are pregnant, breastfeeding, or intend to become pregnant during the course of the study.
17. Individuals ≥ 35 years of age currently using systemic, estrogen-containing contraception or hormone replacement therapy.
18. A positive urine drug screen without evidence of prescribed corresponding concomitant medication(s) at Screening or Day 1.
19. Postpones a decision to quit using tobacco- or nicotine-containing products in order to participate in this study or a previous attempt within (≤) 30 days prior to the signing of the ICF.
20. Drinks more than 21 servings of alcoholic beverages per week or has a positive alcohol breathalyzer result at Screening or Day 1.
21. Employed by a tobacco or nicotine company, the study site, or handles tobacco- or nicotine-containing products as part of their job.
22. Determined by the PI to be inappropriate for this study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2019-11-26 (Actual); Study Completion 2019-11-26 (Actual)

PRIMARY OUTCOMES:
AUECPL 10-240 | 3, 5, 10, 15, 30, 45, 60, 90, 180, and 240 minutes
  Area under the product liking (PL) NRS score-versus-time curve from 10 minutes to 240 minutes after the start of investigational product (IP) use.
Emax PL | 3, 5, 10, 15, 30, 45, 60, 90, 180, and 240 minutes
  Maximum response for product effects with regards to PL score after the start of IP use.
Eoverall IUA | 240 minutes
  Overall intent to use again (IUA), measured at 240 minutes after the start of IP use.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hong, MD, Study Director — RAIS
Locations (2):
- United States (2):
  - New Orleans Center for Clinical Research (NOCCR), Knoxville, Tennessee
  - ICON Clinical Research, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No